CLINICAL TRIAL: NCT07129070
Title: Just-in-Time Training for Youth Mentors: A Strategy for Implementing Evidence-Based Preventive Interventions for Youth in Rural Communities
Brief Title: Just-in-Time Training for Youth Mentors
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Minnesota (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: STUDY00024848
Record Dates: First submitted 2025-07-22; First posted 2025-08-19 (Actual); Last update posted 2026-02-10 (Actual); Status verified 2026-02

CONDITIONS: Mental Health Issue; Depression; Anxiety
MeSH Terms: conditions — Depression; Anxiety Disorders

STUDY DESIGN:
Intervention Model Description: Youth, mentor supervisors, and mentors will be randomized to IPT-AST delivered via JITT-EBP or usual training. Youth will be block randomized using randomly permuted blocks of 2 and 4. Randomization for youth will be stratified by sex and level of depression symptoms (PHQ-9 < 5 and > 5).
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- IPT-AST implemented via Just-In-Time Training (JITT-EBP) (Active Comparator): IPT-AST = Interpersonal Psychotherapy-Adolescent Skills Training
  Interventions: Behavioral: Interpersonal Psychotherapy-Adolescent Skills Training via Just-In-Time Training (JITT) implementation strategy
- IPT-AST implemented via usual training (Active Comparator): IPT-AST = Interpersonal Psychotherapy-Adolescent Skills Training
  Interventions: Behavioral: Interpersonal Psychotherapy-Adolescent Skills Training (IPT-AST) implemented via usual training

INTERVENTIONS:
Behavioral: Interpersonal Psychotherapy-Adolescent Skills Training via Just-In-Time Training (JITT) implementation strategy — IPT-AST is a group-based EBP that aims to prevent depression and support emotional well-being by helping youth develop skills to foster healthy relationships. Youth learn about the links between feelings and interpersonal interactions, and they learn communication strategies and interpersonal problem-solving skills that they can apply to their relationships.
  JITT-EBP integrates (a) self-directed, on-demand, online training modules for mentors and mentor supervisors, (b) synchronous evidence-based supervision strategies, and (c) an apprenticeship delivery model in which EBPs are co-led by an experienced mentor and a novice mentor, providing opportunity for in-the-moment training and support.
  Arms: IPT-AST implemented via Just-In-Time Training (JITT-EBP)
Behavioral: Interpersonal Psychotherapy-Adolescent Skills Training (IPT-AST) implemented via usual training — IPT-AST is a group-based EBP that aims to prevent depression and support emotional well-being by helping youth develop skills to foster healthy relationships. Youth learn about the links between feelings and interpersonal interactions, and they learn communication strategies and interpersonal problem-solving skills that they can apply to their relationships.
  Usual training involves (a) a one-day virtual training conducted by an IPT-AST expert prior to the beginning of the intervention, and (b) synchronous evidence-based supervision strategies.
  Arms: IPT-AST implemented via usual training

SUMMARY:
This study will evaluate the usability, feasibility, and acceptability of a novel multi-level Just-In-Time Training (JITT) implementation strategy (JITT-EBP) that aims to equip mentors and mentor supervisors to implement evidence-based practices (EBPs) with fidelity using methods that are sustainable in rural communities. JITT-EBP integrates (a) self-directed, on-demand, online training modules for mentors and mentor supervisors, (b) synchronous evidence-based supervision strategies, and (c) an apprenticeship delivery model in which EBPs are co-led by an experienced mentor and a novice mentor, providing opportunity for in-the-moment training and support. The study will conduct a pilot hybrid type 2 effectiveness-implementation trial to evaluate the use of JITT-EBP compared to usual training for implementing mentor-delivered Interpersonal Psychotherapy-Adolescent Skills Training (IPT-AST), an evidence-based depression prevention program. 96 adolescents (age 12-17) and their parents, 8-18 mentors (depending on amount of turnover), and 4 mentor supervisors will be enrolled in the trial.

ELIGIBILITY:
Youth and Parent Inclusion Criteria:

* student at a partnering rural middle school or high school
* age 12-17
* have English speaking/reading/writing ability at a level to participate in IPT-AST
* youth's parent has English or Spanish-speaking/reading/writing ability at a level to participate in research activities.

Youth and Parent Exclusion Criteria:

* moderate or severe depression (PHQ-9 > 10)
* active suicidal ideation with a plan and/or intent, requiring higher level of care
* Youth does not have English-speaking ability at a level to participate in IPT-AST
* youth's parent does not have English or Spanish-speaking/reading/writing ability at a level to participate in research activities.

Mentor and Mentor Supervisor Inclusion Criteria:

* age 18 or older
* have completed the typical mentor or mentor supervisor screening and selection process at partnering mentoring organization (including a background check)
* are available to facilitate the program during after-school hours.

Min Age: 12 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 118 (Estimated)
Dates: Start 2025-12-18 (Actual); Primary Completion 2028-04-01 (Estimated); Study Completion 2028-05-31 (Estimated)

PRIMARY OUTCOMES:
Feasibility of Intervention Measure (FIM) - Week 12 | Week 12
  Mentor and mentor supervisor report of JITT-EBP feasibility, with higher value indicating higher feasibility
Acceptability of Intervention Measure (AIM) - Week 12 | Week 12
  youth, parent, mentor, and mentor supervisor report of IPT-AST acceptability, with higher value indicating higher acceptability.
Intervention Appropriateness Measure (IAM) - Week 12 | Week 12
  Mentor and mentor supervisor report of JITT-EBP appropriateness, with higher value indicating higher appropriateness.
Client Satisfaction Questionnaire (CSQ-8) - Week 12 | Week 12
  Youth and parent report of satisfaction with IPT-AST program, with , with higher value indicating more satisfaction.

SECONDARY OUTCOMES:
Fidelity | Week 12
  IPT-AST fidelity checklist
Cost of implementation | Year 2
  Mentor Supervisor hours and hourly wages for recruitment, training, supervision, and IPT-AST delivery. IPT-AST expert hours and hourly wages for training and supervision.
Revised Child Anxiety and Depression Scale-25 (RCADS-25) - Week 6 | Week 6
  25-item scale that measures levels of anxiety and depressed mood. Higher scores indicate higher severity.
Revised Child Anxiety and Depression Scale-25 (RCADS-25) - Week 12 | Week 12
  25-item scale that measures levels of anxiety and depressed mood. Higher scores indicate higher severity.
Revised Child Anxiety and Depression Scale-25 (RCADS-25) - Week 24 | Week 24
  25-item scale that measures levels of anxiety and depressed mood. Higher scores indicate higher severity.
Conflict Behavior Questionnaire-20 (CBQ-20) - Week 6 | Week 6
  A higher score on the CBQ-20 indicates a greater level of conflict in parent-adolescent relationships
Conflict Behavior Questionnaire-20 (CBQ-20) - Week 12 | Week 12
  A higher score on the CBQ-20 indicates a greater level of conflict in parent-adolescent relationships
Conflict Behavior Questionnaire-20 (CBQ-20) - Week 24 | Week 24
  A higher score on the CBQ-20 indicates a greater level of conflict in parent-adolescent relationships
National Survey of Children's Health Social Competence Scale (NSCH-SCS) - Week 6 | Week 6
  A higher score on the NSCH-SCS indicates a higher level of youth social skills, as reported by a parent.
National Survey of Children's Health Social Competence Scale (NSCH-SCS) - Week 12 | Week 12
  A higher score on the NSCH-SCS indicates a higher level of youth social skills, as reported by a parent.
National Survey of Children's Health Social Competence Scale (NSCH-SCS) - Week 24 | Week 24
  A higher score on the NSCH-SCS indicates a higher level of youth social skills, as reported by a parent.
NIH Toolbox -Loneliness Ages 8-17 - Week 6 | Week 6
  A higher score indicates greater severity of loneliness
NIH Toolbox -Loneliness Ages 8-17 - Week 12 | Week 12
  A higher score indicates greater severity of loneliness
NIH Toolbox -Loneliness Ages 8-17 - Week 24 | Week 24
  A higher score indicates greater severity of loneliness
PROMIS Pediatric Item Bank - Peer Relationships - Week 6 | Week 6
  A higher score indicates a more positive experience in relationships with peers
PROMIS Pediatric Item Bank - Peer Relationships - Week 12 | Week 12
  A higher score indicates a more positive experience in relationships with peers
PROMIS Pediatric Item Bank - Peer Relationships - Week 24 | Week 24
  A higher score indicates a more positive experience in relationships with peers
NIH Toolbox - General Life Satisfaction - Week 6 | Week 6
  A higher score indicates more life satisfaction
NIH Toolbox - General Life Satisfaction - Week 12 | Week 12
  A higher score indicates more life satisfaction
NIH Toolbox - General Life Satisfaction - Week 24 | Week 24
  A higher score indicates more life satisfaction
PROMIS Pediatric Short Form v1.0 - Positive Affect - Week 6 | Week 6
  A higher score indicates more positive affect
PROMIS Pediatric Short Form v1.0 - Positive Affect - Week 12 | Week 12
  A higher score indicates more positive affect
PROMIS Pediatric Short Form v1.0 - Positive Affect - Week 24 | Week 24
  A higher score indicates more positive affect
Rosenberg Self-Esteem Scale (RSES) - Week 6 | Week 6
  A higher score indicates higher self-esteem
Rosenberg Self-Esteem Scale (RSES) - Week 12 | Week 12
  A higher score indicates higher self-esteem
Rosenberg Self-Esteem Scale (RSES) - Week 24 | Week 24
  A higher score indicates higher self-esteem

CONTACTS AND LOCATIONS:
Overall Officials: Meredith Gunlicks-Stoessel, PhD, LP, Principal Investigator — University of Minnesota; Lindsey Weiler, PhD, Principal Investigator — University of Minnesota
Locations (1):
- University of Minnesota, Minneapolis, Minnesota, United States

IPD SHARING:
Plan to Share IPD: No